CLINICAL TRIAL: NCT07341581
Title: Supply and Demand-Side Interventions to Improve Uptake of Antenatal Care Services: a Randomized Controlled Trial in Rural Côte d'Ivoire
Brief Title: Improving Uptake of Antenatal Care Services in Rural Côte d'Ivoire
Acronym: Taabo ANC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Tropical & Public Health Institute (Other)
Collaborators: Centre Suisse de Recherches Scientifiques en Cote d'Ivoire (Other); Swiss National Science Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2025-40
Record Dates: First submitted 2025-12-19; First posted 2026-01-14 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Uptake of Antenatal Health Care Services
Keywords: maternal health; sub-Saharan Africa; antenatal care; vouchers; financing

STUDY DESIGN:
Intervention Model Description: This study consists of a randomized controlled experiment with pregnant women. All participants will receive basic antenatal care information through a newly developed introduction video. In addition, participants will be randomly assigned to one of three groups:
  * (1) Control (Information video only for pregnant women)
  * (2) Information video + financial planning for pregnant women only
  * (3) Information video + financial planning for couples together
  Following randomization to a one of the above groups, 10% of women in each group will be randomized to receive vouchers to cover the costs of a set of key antenatal health care services.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- 1a) Information video only (Experimental): Participants in this arm will be shown a short video that describes key recommendations for antenatal care and health during pregnancy, based on national guidelines in Côte d'Ivoire.
  Interventions: Behavioral: Information video
- 1b) Information video + Vouchers (Experimental): Participants in this arm will be shown a short video that describes key recommendations for antenatal care and health during pregnancy, based on national guidelines in Côte d'Ivoire.
  They will also receive vouchers to cover the costs of a set of key antenatal health care services.
  Interventions: Behavioral: Information video; Other: Vouchers
- 2a) Information video + financial planning (Experimental): Participants in this arm will be shown a short video that describes key recommendations for antenatal care and health during pregnancy, based on national guidelines in Côte d'Ivoire.
  They will also receive a financial planning session facilitated by a member of the study team.
  Interventions: Behavioral: Information video; Behavioral: Financial planning session
- 2b) Information video + financial planning + vouchers (Experimental): Participants in this arm will be shown a short video that describes key recommendations for antenatal care and health during pregnancy, based on national guidelines in Côte d'Ivoire.
  They will also receive a financial planning session facilitated by a member of the study team.
  Finally, they will also receive vouchers to cover the costs of a set of key antenatal health care services.
  Interventions: Behavioral: Information video; Behavioral: Financial planning session; Other: Vouchers
- 3a) Information video + financial planning with partners (Experimental): Participants in this arm will be shown a short video that describes key recommendations for antenatal care and health during pregnancy, based on national guidelines in Côte d'Ivoire. They will view it a first time alone, and a second time with their partners.
  They will also receive a financial planning session facilitated by a member of the study team, together with their partners.
  Interventions: Behavioral: Information video; Behavioral: Financial planning session
- 3b) Information video + financial planning with partners + vouchers (Experimental): Participants in this arm will be shown a short video that describes key recommendations for antenatal care and health during pregnancy, based on national guidelines in Côte d'Ivoire. They will view it a first time alone, and a second time with their partners.
  They will also receive a financial planning session facilitated by a member of the study team, together with their partners.
  Finally, they will also receive vouchers to cover the costs of a set of key antenatal health care services.
  Interventions: Behavioral: Information video; Behavioral: Financial planning session; Other: Vouchers

INTERVENTIONS:
Behavioral: Information video — Participants will be shown a short video that describes key recommendations for antenatal care and health during pregnancy, based on national guidelines in Côte d'Ivoire. In arms (1a-1b) and (2a-2b), this video will be shown only to the pregnant woman. In arms (3a-3b), this video will be shown to the pregnant woman together with her partner.
Behavioral: Financial planning session — In this intervention, a member of the study team will facilitate a structured discussion about planning for the expenses of health care services and related transportation costs over the course of pregnancy. The discussion will follow a series of questions and prompts set up as a survey form in ODK (attached to this protocol). The study team member will also share a list of the local prices of recommended antenatal care services. In arms (2a-2b), this intervention is delivered only to pregnant women. In arms (3a-3b), this intervention is delivered to pregnant women together with their partners.
  Arms: 2a) Information video + financial planning; 2b) Information video + financial planning + vouchers; 3a) Information video + financial planning with partners; 3b) Information video + financial planning with partners + vouchers
Other: Vouchers — This intervention consists of vouchers for a pre-defined set of antenatal care services. Pregnant women who are randomized to receive this intervention will be given vouchers for one ultrasound, one "bilan prenatal" (a recommended set of prenatal laboratory tests in Côte d'Ivoire), and a 6-month supply of iron & folic acid supplements (with dosage based on their health care provider's recommendation). The study team will establish agreements with local health facilities to provide services in exchange for these vouchers, with reimbursement by the study team.
  Arms: 1b) Information video + Vouchers; 2b) Information video + financial planning + vouchers; 3b) Information video + financial planning with partners + vouchers

SUMMARY:
The past two decades have brought significant increases in the availability of maternal health care services in many low- and middle-income countries, with a large increase in the number of health facilities that provide these services. However, many women still do not receive the basic services recommended by the World Health Organization. In many settings, antenatal care is associated with substantial financial cost, which means that obtaining high quality care can involve complex intrahousehold bargaining and decision-making. Women have more access to information about these services, but men generally make the financial decisions. If men are unaware of the magnitude and timing of financial needs, securing adequate financial resources may be difficult.

The investigators plan to conduct a randomized-controlled experiment of supply- and demand-side solutions to increase uptake of recommended antenatal care services in rural Côte d'Ivoire, where there are currently substantial gaps in service coverage. Despite Côte d'Ivoire's "free maternity care" policy, many recommended services - including ultrasounds and laboratory tests - continue to carry costs for patients. On the supply side, the study will evaluate the impact of providing key services (including ultrasounds, laboratory testing, and iron and folic acid supplements) for free to pregnant women (in line with Côte d'Ivoire's policy of free provision). On the demand side, the study will evaluate the impact of providing information about antenatal care recommendations to pregnant women (alone or with their partners), and of providing a financial planning session to pregnant women or their partners, or both together. The study will evaluate the impacts of these interventions on the uptake of recommended antenatal care services.

DETAILED DESCRIPTION:
The past two decades have seen significant increases in the uptake of antenatal care (ANC) and facility-based childbirth in low- and middle-income countries (LMICs), driven by expansions in health service availability, reductions in user fees, and introductions of public insurance programs that make services accessible to a larger portion of the population. However, in many cases, expansions in service coverage have not translated into the anticipated improvements in health outcomes.

One of the primary reasons why increases in coverage have not yielded the desired improvements in health outcomes is the low quality of health care services provided in many health facilities in LMICs. These quality gaps appear to be particularly large for women of lower socioeconomic status, who not only tend to attend lower quality health facilities than wealthier or more educated women, but also tend to receive lower quality care within the same health facilities. In many settings, antenatal care is associated with substantial financial cost, which means that obtaining high quality care can involve complex intrahousehold bargaining and decision-making. Women have more access to information about these services, but men generally make the financial decisions. If men are unaware of the magnitude and timing of financial needs, securing adequate financial resources may be difficult.

In Taabo, Côte d'Ivoire, the investigators recently completed a mixed-methods pilot study examining the reasons for gaps in the quality of antenatal care. They found that, while 91% of women attended at least one antenatal care visit, only 44% had the recommended minimum 4 visits. Many also missed out on important recommended services. They found that only 79% of women received at least 1 and only 17% of women received at least 2 ultrasounds over the course of their pregnancies. Only 73% had any laboratory testing (e.g., a blood test to check for anemia). Only 60% reported taking iron and folic acid supplements 30 days per month during their pregnancy. In qualitative interviews, women identified the cost of services as a critical barrier affecting their uptake. Despite Côte d'Ivoire's "free maternity care" policy, many recommended services - including ultrasounds and laboratory tests - continue to carry costs for patients. Qualitative interviews with women raised several potential pathways through which antenatal care service costs could affect uptake. Firstly, in some cases, the services may be unaffordable for some women and their partners. Secondly, a lack of clarity around service prices - particularly in the context of a publicized "free maternity care policy" - makes it challenging for women and their partners to plan for their antenatal care expenditures. Finally, husbands (or male partners) are the main financial decision-makers in many households in the study setting, and they are not always willing to provide resources to cover the costs of antenatal care services.

The investigators plan to conduct a randomized-controlled experiment of supply- and demand-side solutions to increase uptake of recommended antenatal care services. On the supply side, the study will evaluate the impact of providing key services (including ultrasounds, laboratory testing, and iron and folic acid supplements) for free to pregnant women, in line with Côte d'Ivoire's national "free maternity care" policy. On the demand side, the study will evaluate the impact of providing information about antenatal care recommendations to pregnant women (alone or with their partners), and of providing a financial planning session to pregnant women or their partners, or both together. The study will evaluate the impacts of these interventions on the uptake of recommended antenatal care services.

ELIGIBILITY:
Inclusion criteria for pregnant women:

* Currently pregnant
* Aged 15 years or older
* Live in the area served by the Taabo Health & Demographic Surveillance System
* Estimated gestational age of less than 6 completed months of pregnancy

Inclusion criteria for male partners:

* Aged 15 and older
* Married to or currently the main romantic partner of a woman who is enrolled in the study

Min Age: 15 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1290 (Estimated)
Dates: Start 2026-01-16 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Proportion of women receiving recommended antenatal care services | During pregnancy (measured 4-8 weeks after the end of pregnancy)
  The primary endpoint is the proportion of women receiving the following recommended antenatal care services during their pregnancy, as measured through recall during endline surveys with pregnant women:
  * At least four antenatal care visits with a skilled provider AND
  * At least one ultrasound AND
  * At least one laboratory assessment.

SECONDARY OUTCOMES:
Proportion of participants receiving the recommended number of malaria chemoprophylaxis doses during pregnancy | During pregnancy (measured 4-8 weeks after the end of pregnancy)
  Proportion of participants who receive at least three doses of malaria chemoprophylaxis during pregnancy as reported by study participants during endline interviews
Proportion of participants receiving high-quality antenatal care measured using antenatal care booklets | During pregnancy (measured 4-8 weeks after the end of pregnancy)
  High-quality antenatal care (defined as at least 4 antenatal care visits with a skilled provider, at least one ultrasound, and at least one laboratory assessment) as measured through review of antenatal care booklets (as opposed to measurement by maternal recall). This secondary endpoint will only be measured in cases when women have an ANC book available at the time of the endline interview.
Average antenatal care knowledge scores among pregnant women and their partners | Measured 4-8 weeks after the end of pregnancy
  Average scores (among pregnant women and among their partners) on assessments of knowledge of antenatal care recommendations, as measured using the following questions during endline surveys with pregnant women and their partners:
  1. During antenatal care visits, health care providers conduct some examinations and tests. Can you tell me which examinations and tests they should conduct?
  2. During antenatal care visits, health care providers also sometimes give medications or treatments. Can you tell me which medications they should provide to all pregnant women?
  Participants receive 1 point for each correct test or examination they mention in response to Q1 and 1 point for each correct medication or treatment they mention in response to Q2.
Proportion of women who delayed or missed care for financial reasons | Measured 4-8 weeks after the end of pregnancy
  Proportion of women who respond "yes" to one or both of the following questions during endline surveys:
  * During your most recent pregnancy, did you ever delay your visit to the hospital because of financial issues?
  * During your most recent pregnancy, did you ever skip recommended care - like an ultrasound or a blood test - because of money problems?
Proportion of women who are satisfied with the antenatal care health services that they received | Measured 4-8 weeks after the end of pregnancy
  Proportion of women responding "Excellent" or "Very good" to the question, "How would you rate the overall quality of care you received during your most recent pregnancy? Excellent, Very good, Good, Fair, Poor."
Proportion of fathers involved in early care-giving activities | Measured 4-8 weeks after the end of pregnancy
  Proportion of mothers who respond "everyday" or "most days" to the following question during endline surveys: "How often does the father of the child participate in daily care activities such as feeding, bathing, or changing diapers? Every day, most days, some days, or never."
Perinatal mortality as reported by women during endline surveys | Measured 4-8 weeks after the end of pregnancy
  Mortality between 28 weeks of pregnancy and 7 days after birth, as reported by women during endline surveys
Birthweight as reported by women during endline surveys | Measured 4-8 weeks after the end of pregnancy
  Birthweight in grams, as reported by women during endline surveys

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Suisse de Recherches Scientifiques en Cote d'Ivoire, Taabo, Côte d’Ivoire

IPD SHARING:
Plan to Share IPD: Yes
De-identified data files and analytic code will be posted on public repositories at the time of publication of results.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: We plan to share IPD and supporting information at the time of publication.
Access Criteria: IPD and supporting information will be made available on public repositories.